CLINICAL TRIAL: NCT02783495
Title: Feasibility And Efficacy Of An iPad-Based Cognitive Rehabilitation Program In Brain Tumor Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of California, San Francisco (Other)
Collaborators: Tilburg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16106; NCI-2017-01881 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2016-05-22; First posted 2016-05-26 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Glioma
Keywords: glioma; neurocognitive; quality of life
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device: iPad (Experimental): Patients with brain tumors receive an iPad with the ReMind app. The patients will use the app to train neurocognitive and compensatory skills for 3 hours per week over the course of 12 weeks (36 hours in total)
  Interventions: Behavioral: Device: iPad

INTERVENTIONS:
Behavioral: Device: iPad — All patients will receive baseline neurocognitive and quality of life testing, followed by 3 months of the iPad-based intervention. At the end of the baseline visit, subjects will be lent an iPad to take home (or will be assisted in the installation of the ReMind app on their personal iPad) and instructed in the use of the ReMind app (and more basic iPad skills, if necessary). Subjects will review the intervention schedule (approximately 3 hours per week). Testing will be repeated 3 months after the baseline visit (i.e., immediately after the intervention) and 9 months after the baseline visit (i.e., 6 months after completion of the intervention), both time-points including a new MRI.

SUMMARY:
This pilot clinical trial studies how well an iPad-based cognitive rehabilitation program works in improving quality of life in patients with grade II-III glioma. An iPad-based cognitive rehabilitation program may help to increase patients cognitive function and quality of life, and may provide doctors with valuable information for optimizing care of patients with brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed WHO grade 2 or 3 gliomas.
* Patients must be > 18 years old
* Patients must have a life expectancy > 12 weeks.
* Patients must have a Karnofsky performance status of > 70.
* This study was designed to include women and minorities, but was not designed to measure differences between them. Males and females will be recruited with no preference to gender. Minorities will actively be recruited to participate. No exclusion to this study will be based on race.
* Patients must speak and be able to read English fluently.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must sign an authorization for the release of their protected health information.
* Patients may not be known to be HIV-positive. HIV testing is not required for study participation.
* Patients must not have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
* Patients must be receiving MRI scans at UCSF
* Patients must be clinically stable and off treatment (e.g. radiation or chemotherapy) for ≥ 6 months
* Patients must be ≥ 6 months from craniotomy
* Patients must have subjective complaints of cognitive deficits.
* Patients must have adequate seizure control and be on a stable, or decreasing, dose of anti-epileptics

Exclusion Criteria:

* Patients who are not able to comply with study and/or follow-up procedures.
* Patients who do not have home access to the Internet.
* Patients who, based on the physician's opinion, are unable to participate in neurocognitive testing and/or neurocognitive rehab secondary to significant neurologic deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects who complete the intervention | At 3 months after start of training
  Subjects who complete all of the intervention exercises (approximately 36 hours of intervention).
Patient-reported ease of use | At 3 months after start of training
  Questionnaire based measure of ease of use as a measure of feasibility.
Patient-reported user satisfaction | At 3 months after start of training
  Questionnaire based measure of user satisfaction as a measure of feasibility.
Change in attention | At baseline, 3 months past training start, 9 months past training start
  Evaluation of visual attention on the NIH Toolbox Flanker Inhibitory Control and Attention Test. The attention score ranges from 0 to 10 (10 = best performance)
Change in working memory | At baseline, 3 months past training start, 9 months past training start
  Evaluation of working memory using the NIH Toolbox List Sorting Working Memory Test. Higher scores on each of these indicate higher levels of working memory.
Change in Quality of Life | At baseline, 3 months past training start, 9 months past training start
  Measurement of general quality of life (QOL) using Functional Assessment of Cancer Therapy-Brain (FACT-Br), a multi-item questionnaire. Higher ratings suggest higher QOL.

SECONDARY OUTCOMES:
Improvement on neurocognitive testing | At baseline, 3 months past training start, 9 months past training start
  Improvement on neurocognitive testing as measured by the NIH Toolbox assessment after the intervention.
Subjective assessment of cognitive symptoms will be assessed | At baseline, 3 months past training start, 9 months past training start
  Subjective assessment of cognitive symptoms using the Functional Assessment of Cancer Therapy: Cognitive Function (FACT-Cog) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jennie W Taylor, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Subject data collected or generated as the result of participation in this study may be shared with co-investigators at the Tilburg University, The Netherlands, who developed the ReMind application. This may include clinical data, pathology data, imaging data, image files, and neurocognitive assessment results. All such data will be identified only by the subject's study code. All clinical research staff from The Netherlands will maintain all study materials in compliance with applicable laws, regulations and policies.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: July 2016- May 2019